CLINICAL TRIAL: NCT01625208
Title: Standard Supraclavicular Block Versus Low-Volume Supraclavicular Block Plus Ulnar or Median Nerve Block for Hand Surgery in the Ulnar or Median Nerve Distribution
Brief Title: Supraclavicular Versus Combined Block for Ulnar and Median Distribution Hand Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00027213
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2015-04

CONDITIONS: Hand Surgery (Ulnar or Median Distribution); Peripheral Nerve Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combined nerve block (Experimental): Participants in this group will receive a supraclavicular brachial plexus block plus a median or ulnar nerve block.
  Interventions: Procedure: Combined nerve block
- Single nerve block (Active Comparator): Participants in this group will receive a supraclavicular brachial plexus block only.
  Interventions: Procedure: Supraclavicular block

INTERVENTIONS:
Procedure: Combined nerve block — Combined supraclavicular brachial plexus block plus ulnar or median nerve block (depending on the location of surgery)
  Arms: Combined nerve block
Procedure: Supraclavicular block — Standard supraclavicular brachial plexus block
  Arms: Single nerve block

SUMMARY:
This study will examine how successfully nerves are blocked or frozen for hand surgery. Traditionally, the nerves are frozen at the base of the neck, just above the clavicle or collarbone (the supraclavicular block). This is mostly successful by itself, and provides anesthesia of the entire arm. Occasionally, an additional nerve block is required further down the arm, as the supraclavicular block may have missed a segment, or it is taking too long to come on. In this study the investigators will compare the traditional technique, with a similar but lower volume supraclavicular block plus an immediate low volume block of one nerve further down the arm (the ulnar or median nerve block, depending on which digits are being operated on). The investigators will compare success rates, speed of onset, procedural comfort and length of time of weakness and numbness, plus any adverse events.

DETAILED DESCRIPTION:
Background

Regional anesthesia is commonly employed for surgery on the hand. It is well tolerated by most patients and has a high safety record.

The most common form of regional anesthesia for this surgery is the supraclavicular block which is successful in most cases. Occasionally an additional nerve block and/or moderate sedation is required. The most frequent additional nerve blocks required are for the ulnar and median nerves.

This study aims to address whether a low volume supraclavicular block plus a selective ulnar or median nerve block reduces the time taken for onset of anesthesia, reduces the time of post-operative complete limb immobility, improves the surgical success of the block, and increases patient satisfaction, compared to a standard block.

The study will be powered to detect a 25% difference in successful surgical anesthesia.

Purpose

To ascertain whether the addition of an ulnar or median nerve block to a lower volume supraclavicular block speeds up the onset and consistency of anesthesia, and the return of limb function in patients undergoing hand surgery when compared to a standard supraclavicular block.

Hypothesis

Low volume supraclavicular block plus selective distal nerve blocks will speed up the onset of anesthesia, improve surgical anesthetic success and decrease the time to the return of upper limb function when compared to a standard supraclavicular block.

Study population

Patients over 18 years of age, listed for hand surgery in the ulnar or median distribution at the University of Alberta Hospital. The study will commence following ethical approval and will run until 160 patients are enrolled.

Exclusion criteria

* Patient refusal
* Allergy to amide local anesthetics
* Severe coagulopathy
* Bilateral upper limb surgery
* Surgery involving bone graft from the iliac crest
* Request for general anesthetic from surgical or research team (for example, nerve stimulation studies)

Methods

Consent will be obtained by one of the investigators. Patients not wishing to participate in the study will receive either a brachial plexus block or a general anesthetic as deemed appropriate by the attending anesthesiologist.

Patients to undergo surgery on the ring or pinky fingers will be randomised to receive either a standard supraclavicular block, or a low volume supraclavicular block plus ulnar nerve block. Patients receiving surgery on the thumb, index, or middle fingers will be randomized in a similar fashion to a separate "median" group. All blocks will be placed in a designated block area prior to transfer to the operating room by either an experienced staff anesthesiologist or a supervised fellow in regional anesthesia. The block will be assessed prior to surgery for motor and sensory dysfunction, and the block may be augmented if necessary. The surgeon will determine the effectiveness of the surgical anesthesia, and will indicate a need for surgical local anesthetic top up, heavy sedation or general anesthesia to the anesthesiologist. Sedation can also be administered as per patient request.

Post-operatively, a patient satisfaction questionnaire will be completed. A phone call will be conducted the following day.

Primary outcome measures

1. Successful surgical anesthesia

Secondary outcome measures

1. Time to successful anesthetic block
2. Procedural time
3. Duration of analgesia
4. Duration of weakness
5. Patient satisfaction

Safety concerns

Ultrasound-guided supraclavicular blocks have been performed for many years, with a low complication rate. The addition of a peripheral nerve block is not uncommon, and poses minimal additional risk.

Major concerns

1. Pneumothorax
2. Nerve damage
3. Intravascular injection causing local anesthetic toxicity
4. Infection

Minor concerns

1. Block failure
2. Transient hemidiaphragmatic paresis
3. Transient Horner's syndrome
4. Transient recurrent laryngeal nerve palsy
5. Haematoma at injection site

Study Protocol

Patients will be transferred to the block area. Midazolam will be titrated to an appropriate level. A time out procedure will be undertaken to ensure the correct side is being blocked. The skin will be disinfected. The ultrasound probe will scan the supraclavicular fossa to identify the subclavian artery. The brachial plexus is identified postero-lateral to the artery.

Standard supraclavicular block

The skin will be infiltrated with lidocaine. A needle attached to a nerve stimulator will be introduced. The target will be an area infero-medial to the brachial plexus. In this position 10 - 20 ml of a 3:1 Lidocaine 2%: 0.5% Bupivacaine solution is injected. A more superficial injection is then made. A further 10-20 mls of the Lidocaine:Bupivacaine solution is deposited. The total volume will be recorded with a maximum of 30mls.

Low volume supraclavicular block with ulnar nerve block

The skin infiltration and target of the needle is the same as for the standard supraclavicular block. However, a maximum of 15ml of the solution will be injected. The arm is then abducted and supinated. The ulnar artery is identified. The ulnar nerve is seen medial to the artery. 5ml of the solution is deposited adjacent to the nerve.

Low volume supraclavicular block with median nerve block

The skin infiltration and target of the needle is the same as for the standard supraclavicular block. However, a maximum of 15ml of the solution will be injected. The patient's elbow is flexed and the nerve is visualized on ultrasound in the antecubital fossa lying medial to the brachial artery. Anesthetic solution is deposited in the forearm to target the median nerve.

Intra-operative management

Following block assessment, the patient will be transferred to the operating theatre. Additional midazolam may be given. Propofol at 50mcg/kg/minute will be commenced if required, and the rate can be increased to 75mcg/kg/minute. If the patient is unable to tolerate the procedure, sedation can be increased to at least 100mcg/kg/minute and the block is deemed an unsuccessful surgical block.

Block Assessment

Patients will be assessed for sensory and motor blockade of each nerve at 5 minute intervals.

A successful anesthetic block will be defined as a sensation score in the ulnar or median area of 0 or 1, and an ulnar or median motor score of 2 or less. If this does not occur in the standard group, an ulnar or median nerve block will be performed. If this does not occur in the combined group, a general anesthetic will occur.

Nerve block extent may also be assessed by objective means (e.g., strength testing with a dynamometer).

A successful surgical block will be defined as requiring no further LA top-up or infiltration, and sedation no greater than 75mcg/kg/min.

Data collection

Data will be collected on a study sheet. Information will be kept confidential and there will be no patient identifiers on the form.

The data collected will be age, sex, height and weight, the type of block used, the amount of local anesthetic used, the length of time taken to perform all blocks, the block assessment data. Intraoperative data will note whether additional local anaesthetic, heavy sedation or general anesthesia was required and the reason. Post-operative data will be a patient questionnaire asking about block-related and surgery-related pain score. A follow up phone call the day after surgery will determine the timing of return of power and sensation of the arm.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Surgery on distal upper extremity amenable to a regional anesthetic involving the ulnar (ring, pinky fingers) or median (thumb, index, middle fingers) distribution.

Exclusion Criteria:

* Patient refusal
* Allergy to amide local anesthetics
* Severe coagulopathy
* Bilateral upper limb surgery
* Surgery involving bone graft from the iliac crest
* Request for general anesthetic from surgical or research team (for example, nerve stimulation studies)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2013-02 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Successful anesthesia, defined as no additional local anesthetic or heavy sedation required. | From injection of local anesthetic to suitable nerve blockade for surgery; approximately 20 minutes
  Successful anesthesia will be determined by assessing the nerve block(s) following injection of local anesthetic, and deeming the block sufficient enough for surgery to proceed without any need for additional local anesthetic or heavy sedation. The period between the initial injection and successful anesthesia is approximately 20 minutes, depending on the patient.

SECONDARY OUTCOMES:
Time to successful anesthetic block from withdrawal of final needle | Approximately 20 minutes
  The period between final withdrawal of the needle to successful nerve block following assessment will be timed.
Time for procedure, from placement of probe on skin to withdrawal of needle | Approximately 30 minutes
  The period between initial placement and positioning of the ultrasound probe on the patient to final withdrawal of the needle will be timed.
Duration of analgesia | Approximately 6 hours
  The length of time between successful nerve block (i.e., when patient is ready for surgery) to the time the anesthesia wears off will be sought.
Duration of motor blockade | Approximately one hour
  The time taken for the patient to recover motor capability in the area anesthetized following local anesthetic injection will be determined.
Patient satisfaction | 24-48 hours
  Patient satisfaction with reduction of pain and recovery of motor capability will be assessed in the 24-48 hour period following surgery.

CONTACTS AND LOCATIONS:
Overall Officials: James Cameron, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] McCartney CJ, Brull R, Chan VW, Katz J, Abbas S, Graham B, Nova H, Rawson R, Anastakis DJ, von Schroeder H. Early but no long-term benefit of regional compared with general anesthesia for ambulatory hand surgery. Anesthesiology. 2004 Aug;101(2):461-7. doi: 10.1097/00000542-200408000-00028. PMID 15277930
- [Background] Perlas A, Lobo G, Lo N, Brull R, Chan VW, Karkhanis R. Ultrasound-guided supraclavicular block: outcome of 510 consecutive cases. Reg Anesth Pain Med. 2009 Mar-Apr;34(2):171-6. doi: 10.1097/AAP.0b013e31819a3f81. PMID 19282715
- [Background] Kapral S, Krafft P, Eibenberger K, Fitzgerald R, Gosch M, Weinstabl C. Ultrasound-guided supraclavicular approach for regional anesthesia of the brachial plexus. Anesth Analg. 1994 Mar;78(3):507-13. doi: 10.1213/00000539-199403000-00016. PMID 8109769
- [Background] Duggan E, El Beheiry H, Perlas A, Lupu M, Nuica A, Chan VW, Brull R. Minimum effective volume of local anesthetic for ultrasound-guided supraclavicular brachial plexus block. Reg Anesth Pain Med. 2009 May-Jun;34(3):215-8. doi: 10.1097/AAP.0b013e31819a9542. PMID 19587618
- [Background] Fredrickson MJ, Ting FS, Chinchanwala S, Boland MR. Concomitant infraclavicular plus distal median, radial, and ulnar nerve blockade accelerates upper extremity anaesthesia and improves block consistency compared with infraclavicular block alone. Br J Anaesth. 2011 Aug;107(2):236-42. doi: 10.1093/bja/aer101. Epub 2011 May 15. PMID 21576095
- [Background] Hadzic A, Dilberovic F, Shah S, Kulenovic A, Kapur E, Zaciragic A, Cosovic E, Vuckovic I, Divanovic KA, Mornjakovic Z, Thys DM, Santos AC. Combination of intraneural injection and high injection pressure leads to fascicular injury and neurologic deficits in dogs. Reg Anesth Pain Med. 2004 Sep-Oct;29(5):417-23. doi: 10.1016/j.rapm.2004.06.002. PMID 15372385
- [Background] Fredrickson MJ, Patel A, Young S, Chinchanwala S. Speed of onset of 'corner pocket supraclavicular' and infraclavicular ultrasound guided brachial plexus block: a randomised observer-blinded comparison. Anaesthesia. 2009 Jul;64(7):738-44. doi: 10.1111/j.1365-2044.2009.05918.x. PMID 19624628